CLINICAL TRIAL: NCT05442879
Title: The Effects of a Knowledge Translation Intervention With an ACL Prevention Program on Implementation, Injury Rates, and Performance in Youth Soccer Players
Brief Title: Knowledge Translation Intervention for ACL Injury Prevention Program in Youth Soccer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Community Foundation of Greater Flint (Unknown)
Responsible Party: Principal Investigator, William Suits, Assistant Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00214282
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Anterior Cruciate Ligament Injuries; Lower Extremity Problem
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knowledge Translation Intervention (Experimental): The group participating in the KT intervention program will participate in focus groups, individual meetings, and receive videos, informational handouts and on-field training from the researchers. The researchers and participants will work together to determine barriers and facilitators towards implementation of an ACL-IPP, and create an ACL-IPP that follows established clinical practice guidelines and is individualized to the local contextual needs.
  Interventions: Behavioral: Knowledge Translation Intervention
- Educational Handout (Active Comparator): The coaches will receive an educational handout describing an ACL-IPP.
  Interventions: Behavioral: Educational handout

INTERVENTIONS:
Behavioral: Knowledge Translation Intervention — The KT intervention utilizes the communications between the teams and the researchers to promote implementation of the ACL-IPPs. The meetings will provide opportunities for mutually beneficial learning from the researchers, and feedback from the coaches on how to best implement strategies through local barriers in order to facilitate necessary changes to promote ACL-IPP usage while adhering to clinical practice guideline recommendations.
  Arms: Knowledge Translation Intervention
Behavioral: Educational handout — Educational handout describing a commonly cited ACL-IPP.
  Arms: Educational Handout

SUMMARY:
Anterior cruciate ligament (ACL) injuries of the knee are common in youth soccer players, and show an even higher prevalence in female soccer players. Clinical practice guidelines recommend ACL injury prevention programs (ACL-IPP) to reduce injury risk, yet implementation in amateur youth soccer is low, reducing actual real-world effectiveness. This trial is a pragmatic effectiveness trial for ACL injury prevention for amateur youth soccer players, using a knowledge translation intervention with the Knowledge-to-Action Framework.

DETAILED DESCRIPTION:
ACL injury prevention programs (ACL-IPP) are exercise programs recommended by clinical practice guidelines that have been shown to reduce the risk of an ACL injury. However, implementation of these programs is low, which reduces the real-world effectiveness of these programs. This project will assess a knowledge translation intervention with youth soccer programs for implementation of ACL-IPPs utilizing the Knowledge-to-Action Framework. The main educational intervention will be a knowledge translation (KT) intervention between the researchers, and coaches/players of youth soccer programs within the state of Michigan. Specifics of the knowledge translation intervention will or may include focus groups, surveys, in-person training, video handouts, and paper handouts. This will be compared to coaches/teams that are offered a handout that describes an evidence-based ACL-IPP.

ELIGIBILITY:
Inclusion Criteria:

* Amateur youth soccer organizations within southern Michigan.

Exclusion Criteria:

* Players above the age of 19 or below the age of 14
* Teams that have dedicated medical staffing

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 671 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Uptake of ACL-IPP | up to 2 years
  Reported frequency of implementation of ACL-IPP
Number of ACL injuries | up to 2 years

SECONDARY OUTCOMES:
Change in 5-10-5 test time | 2-4 months
  Average change in 5-10-5 (Pro Agility) test time
Change in horizontal jump distance | 2-4 months
  Average change in forward jumping distance
Change in 10 meter forward run time | 2-4 months
  Average change in time spent running 10 meters
Number of time-loss lower extremity injuries | up to 2 years
  Number of reported injuries to the foot, ankle, knee, and hip which cause a player to miss time with team

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan-Flint, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided